CLINICAL TRIAL: NCT00610545
Title: Atorvastatin 80mg Versus Atorvastatin 20mg in Perioperative Vascular Surgery to Evaluate Cardiovascular Outcomes
Brief Title: Atorvastatin in Perioperative Vascular Surgery - Pilot Study
Acronym: APVS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: RAITANY COSTA DE ALMEIDA, STATE UNIVERSITY OF CAMPINAS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FCM-UNICAMP - 620/2006; 0492.0.146.000-06
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Vascular Surgery
Keywords: ATORVASTATIN; VASCULAR SURGERY; CARDIOVASCULAR OUTCOMES
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Use Atorvastatin 80mg for 60 days , and the vascular surgery will be made between day-7 and day-60
  Interventions: Drug: Atorvastatin
- 2 (Active Comparator): Use Atorvastatin 20 mg for 60 days , and the vascular surgery will be made between day-7 and day-60
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80 mg; Use Atorvastatin for 60 days , and the vascular surgery will be made between day-7 and day-60
  Arms: 1
Drug: Atorvastatin — Atorvastatin 20 mg; Use Atorvastatin for 60 days , and the vascular surgery will be made between day-7 and day-60
  Arms: 2

SUMMARY:
This study is designed to determine if the use of atorvastatin (Lipitor), a member of the HMG coA reductase inhibitor class of drugs referred to as statins, will reduce cardiovascular outcomes ( mortality - myocardial infarction - stroke ) when given in high doses in comparative standard doses in the perioperative period of major vascular surgery.

Abdominal aortic aneurysm , Carotid endarterectomy , Revascularization of lower limbs

ELIGIBILITY:
Inclusion Criteria:

* Vascular surgery (abdominal aortic aneurysm , carotid endarterectomy , limbs revascularization)

Exclusion Criteria:

* Pregnant or lactating women
* Patient with sensitivity to atorvastatin
* Patient has elevations in certain laboratory values (CK, AST, ALT)
* Known history of active hepatic disease or known hepatic insufficiency
* Patients participating in another clinical trial
* Prior statin therapy to include: >10 mg of atorvastatin (Lipitor) or >20 mg of other HMG-CoA Reductase Inhibitors (statins) or use rosuvastatin
* Serious infectious disease after surgery
* Known history of cancer

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
mortality ; myocardial infarction ; stroke | within 90 days after surgery

SECONDARY OUTCOMES:
Change and percent change from baseline to the surgery of treatment for LDL-C, HDL-C, TC, and TG for subjects | within 24h before surgery
Change and percent change from baseline to the surgery of treatment for hs-CRP | within 24h before surgery
Safety of atorvastatin through laboratory assessment | within 24h before surgery

CONTACTS AND LOCATIONS:
Overall Officials: OTAVIO COELHO, PhD, Study Director — STATE UNIVERSITY CAMPINAS; RAITANY C ALMEIDA, MD, Principal Investigator — STATE UNIVERSITY CAMPINAS
Locations (1):
- Clinics Hospital - State University Campinas, Campinas, São Paulo, Brazil